CLINICAL TRIAL: NCT01987011
Title: Randomized, Double Blind, Multicenter, Phase III Study to Evaluate the Immunogenicity and Safety of 'MG1109(Egg-based, Pre-pandemic Influenza(H5N1) Vaccine)' Administered Intramuscularly in Healthy Adult Volunteers
Brief Title: Phase III Study to Evaluate the Immunogenicity and Safety of MG1109 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MG1109_P3
Record Dates: First submitted 2013-07-22; First posted 2013-11-19 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Influenza
Keywords: Avian influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MG1109 (Experimental): MG1109 0.5 mL Intramuscularly injection, twice at an interval of 21 days
  Interventions: Biological: MG1109
- Placebo (Placebo Comparator): Placebo(for MG1109) 0.5 mL Intramuscularly injection, twice at an interval of 21 days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MG1109
  Arms: MG1109
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the investigational vaccine in the subjects during their participation in the study.

DETAILED DESCRIPTION:
MG1109 is purified, inactivated influenza viral antigen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are available for follow-up during the study

Exclusion Criteria:

* Subjects with history of exposure to the H5N1 subtype or H5N1 subtype vaccine
* Subjects with immune system disorder including immune deficiency disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving post-vaccination Hemagglutination Inhibition(HI) antibody titer ≥ 1:40 | 1st vaccination ~ 21 days after 2nd vaccination
Percentage of subjects achieving post-vaccination seroconversion for Hemagglutination Inhibition(HI) antibody | 1st vaccination ~ 21 days after 2nd vaccination
GMR(Geometric Mean Ratio) of Hemagglutination Inhibition(HI) antibody titer at post-vaccination compared to pre-vaccination | 1st vaccination ~ 21 days after 2nd vaccination
The percentage of subjects reporting solicited adverse events from the date of vaccination until 7 days after each vaccination | Each vaccination ~ 7 days after each vaccination
The percentage of subjects reporting unsolicited adverse events from the date of 1st vaccination until 24weeks after 2nd vaccination | 1st vaccination ~ 24 weeks after 2nd vaccination

SECONDARY OUTCOMES:
GMT(Geometric Mean Titer) of Hemagglutination Inhibition(HI) antibody titer pre-vaccination and post-vaccination | 1st vaccination ~ 21 days after 2nd vaccination
GMT(Geometric Mean Titer) and GMR(Geometric Mean Ratio) of neutralizing antibody titer pre-vaccination and post-vaccination | 1st vaccination ~ 21 days after 2nd vaccination
Vital signs(body temperature, pulse) | 1st vaccination ~ 21 days after 2nd vaccination
The results of physical examinations | 1st vaccination ~ 21 days after 2nd vaccination
Lab results(Hematology, Blood chemistry, Urinalysis) | 1st vaccination ~ 21 days after 2nd vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, MD, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (4):
- South Korea (4):
  - Korea University Ansan Hospital, Ansan
  - Inha University Hospital, Inchon
  - Korea University Guro Hospital, Seoul
  - Catholic University Of Korea ST. Vincent's Hospital, Suwon